CLINICAL TRIAL: NCT01892371
Title: Phase I/II Study of the Combination of Quizartinib (AC220) With 5-Azacytidine or Low-Dose Cytarabine for the Treatment of Patients With Acute Myeloid Leukemia (AML) and Myelodysplastic Syndrome (MDS)
Brief Title: Quizartinib With Azacitidine or Cytarabine in Treating Patients With Relapsed or Refractory Acute Myeloid Leukemia or Myelodysplastic Syndrome
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2012-1047; NCI-2018-01813 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2012-1047 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2013-07-01; First posted 2013-07-04 (Estimated); Results first posted 2024-02-28 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2024-10

CONDITIONS: FLT3 Gene Mutation Negative; FLT3 Internal Tandem Duplication Positive; Recurrent Acute Myeloid Leukemia; Recurrent Chronic Myelomonocytic Leukemia; Recurrent Myelodysplastic Syndrome; Refractory Acute Myeloid Leukemia; Refractory Chronic Myelomonocytic Leukemia; Refractory Myelodysplastic Syndrome
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Leukemia, Myelomonocytic, Chronic; Myelodysplastic Syndromes | interventions — Azacitidine; Cytarabine; quizartinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Phase 1 Arm I (quizartinib, azacitidine) (Experimental): Patients receive quizartinib PO QD on days 5-28 of cycle 1 and on days 1-28 of subsequent cycles and azacitidine SC or IV over 10-40 minutes on days 1-7. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Azacitidine; Drug: Quizartinib
- Phase 1 Arm II (quizartinib, cytarabine) (Experimental): Patients receive quizartinib PO QD on days 5-28 of cycle 1 and on days 1-28 of subsequent cycles and cytarabine SC BID on days 1-10. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Cytarabine; Drug: Quizartinib
- Phase 2 Arm I (quizartinib, azacitidine) (Experimental): Patients receive quizartinib PO QD on days 5-28 of cycle 1 and on days 1-28 of subsequent cycles and azacitidine SC or IV over 10-40 minutes on days 1-7. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Azacitidine; Drug: Quizartinib
- Phase 2 Arm II (quizartinib, cytarabine) (Experimental): Patients receive quizartinib PO QD on days 5-28 of cycle 1 and on days 1-28 of subsequent cycles and cytarabine SC BID on days 1-10. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Cytarabine

INTERVENTIONS:
Drug: Azacitidine — Given SC or IV
  Other Names: 5 AZC; 5-AC; 5-Azacytidine; 5-AZC; Azacytidine; Azacytidine, 5-; Ladakamycin; Mylosar; U-18496; Vidaza
  Arms: Phase 1 Arm I (quizartinib, azacitidine); Phase 2 Arm I (quizartinib, azacitidine)
Drug: Cytarabine — Given SC
  Other Names: .beta.-Cytosine arabinoside; 1-.beta.-D-Arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-.beta.-D-Arabinofuranosylcytosine; 1-Beta-D-arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-Beta-D-arabinofuranosylcytosine; 1.beta.-D-Arabinofuranosylcytosine; 2(1H)-Pyrimidinone, 4-Amino-1-beta-D-arabinofuranosyl-; 2(1H)-Pyrimidinone, 4-amino-1.beta.-D-arabinofuranosyl-; Alexan; Ara-C; ARA-cell; Arabine; Arabinofuranosylcytosine; Arabinosylcytosine; Aracytidine; Aracytin; Aracytine; Beta-Cytosine Arabinoside; CHX-3311; Cytarabinum; Cytarbel; Cytosar; Cytosine Arabinoside; Cytosine-.beta.-arabinoside; Cytosine-beta-arabinoside; Erpalfa; Starasid; Tarabine PFS; U 19920; U-19920; Udicil; WR-28453
  Arms: Phase 1 Arm II (quizartinib, cytarabine); Phase 2 Arm II (quizartinib, cytarabine)
Drug: Quizartinib — Given PO
  Other Names: AC-220; AC010220; AC220
  Arms: Phase 1 Arm I (quizartinib, azacitidine); Phase 1 Arm II (quizartinib, cytarabine); Phase 2 Arm I (quizartinib, azacitidine)

SUMMARY:
This phase I/II trial studies the side effects and best dose of quizartinib when given in combination with azacitidine or cytarabine in treating patients with acute myeloid leukemia or myelodysplastic syndrome that have come back (relapsed) or are not responding to treatment (refractory). Quizartinib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as azacitidine and cytarabine work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving quizartinib with azacitidine or cytarabine may work better in patients with acute myeloid leukemia or myelodysplastic syndrome.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the dose limiting toxicity (DLT) and maximum tolerated dose (MTD) of the combination of quizartinib (AC220) with either azacitidine (5-azacitidine [AZA]) or low-dose cytarabine (LDAC) in patients with acute myeloid leukemia (AML) or high-risk myelodysplastic syndrome (MDS). (Phase I) II. To determine the clinical activity of the combination of quizartinib with either AZA or LDAC in patients with AML or MDS. (Phase II)

SECONDARY OBJECTIVES:

I. To determine the clinical activity of the combination of quizartinib with either AZA or LDAC in patients with AML or MDS. (Phase I) II. To determine the safety of the combination of quizartinib with either AZA or LDAC in patients with AML or MDS. (Phase II) III. To determine the induction of hypomethylation, deoxyribonucleic acid (DNA) damage and FLT3 signaling during therapy with this combination and its correlation with response. (Phase I and II) IV. To determine the effect of this combination therapy on plasma levels of FLT3-ligand. (Phase I and II) V. To determine the pharmacodynamics of this combination therapy in patients with AML or high-risk MDS. (Phase I and II)

OUTLINE: This is a phase I, dose-escalation study of quizartinib followed by a phase II study. Participants are assigned to 1 of 2 arms.

ARM I: Patients receive quizartinib orally (PO) once daily (QD) on days 5-28 of cycle 1 and on days 1-28 of subsequent cycles and azacitidine subcutaneously (SC) or intravenously (IV) over 10-40 minutes on days 1-7. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

ARM II: Patients receive quizartinib PO QD on days 5-28 of cycle 1 and on days 1-28 of subsequent cycles and cytarabine SC twice daily (BID) on days 1-10. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 6-12 months.

ELIGIBILITY:
Inclusion Criteria:

* PHASE I
* Refractory or relapsed disease defined as follows: patients with MDS or chronic myelomonocytic leukemia (CMML) should have failed prior therapy (e.g., with a hypomethylating agent, clofarabine, and/or with lenalidomide); patients with AML should have failed any prior induction therapy or have relapsed after prior therapy; patients (any age) with MDS or CMML who received therapy with a hypomethylating agent and progress to AML are eligible at the time of diagnosis of AML regardless any prior therapy for AML. The World Health Organization (WHO) classification will be used for AML; patients with any of the eligible diagnoses who have received no prior therapy are eligible if not candidates to receive standard intensive therapy (i.e., high-dose cytarabine-based chemotherapy).
* Patients are eligible regardless of their FLT3 mutation status.
* PHASE II
* COHORT 2A: Patients with MDS, CMML or AML who are either: age 60 years or older and newly diagnosed, previously untreated. Prior therapy with hydroxyurea or single agent ara-C for the purpose of control of white blood cells (WBC) is acceptable.; age 18 years or older and with refractory or relapse disease who have received no more than one prior treatment regimen and will be receiving first salvage. For this purpose, a second induction cycle with the same drugs used during the first cycle, consolidation chemotherapy or stem cell transplant in complete remission (CR) (or complete response with incomplete platelet recovery [CRp] or complete response with incomplete bone marrow recovery [CRi]) will be considered part of the prior regimen. Prior therapy for MDS (or other malignancies) is not considered a prior regimen for AML in patients who progress from MDS (or other malignancies).
* COHORT 2A: Patients (any age) with MDS or CMML who received therapy with a hypomethylating agent and progress to AML are eligible at the time of diagnosis of AML regardless any prior therapy for AML. The WHO classification will be used for AML.
* COHORT 2A: Patients must have evidence of FLT3 ITD in their most recent assessment.
* COHORT 2B: Patients with MDS, CMML or AML who are either: Age 60 years or older and newly diagnosed, previously untreated. Prior therapy with hydroxyurea or single agent ara-C for the purpose of control of WBC is acceptable or age 18 years or older and with refractory or relapse disease who have received no more than two prior treatment regimens and will be receiving second salvage, or who have received a prior SCT and will be receiving their first salvage. For this purposes, a second induction cycle with the same drugs used during the first cycle, consolidation chemotherapy or stem cell transplant in CR (or CRp or CRi) will be considered part of the prior regimen. Prior therapy for MDS (or other malignancies) is not considered a prior regimen for AML in patients who progress from MDS (or other malignancies)
* COHORT 2B: Patients (any age) with MDS or CMML who received therapy with a hypomethylating agent and progress to AML are eligible at the time of diagnosis of AML regardless any prior therapy for AML. The WHO classification will be used for AML
* COHORT 2B: Patients must have no evidence of FLT3 mutations in their most recent assessment
* PHASE I AND II
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2.
* Bilirubin =< 2 x upper limit of normal (ULN).
* Alanine aminotransferase (ALT) =< 2.5 x ULN.

  * For patients with suspected liver infiltration from leukemia ALT should be =< 5 ULN.
* Creatinine =< 2 x ULN.
* Serum potassium, magnesium, and calcium (normalized for albumin) levels should be at least within institutional normal limits.
* Patients must provide written informed consent.
* Patients must have been off chemotherapy for 2 weeks prior to entering this study, unless there is evidence of rapidly progressive disease, and must have recovered from the toxic effects of that therapy to at least grade 1. Use of hydroxyurea for patients with rapidly proliferative disease is allowed before the start of study therapy and for the first four weeks on therapy. The additional days of hydrea after 28 is permitted as clinically indicated, on case by case basis after discussion with the principal investigator (PI). Other agents given transiently with the intention to control rapid proliferation such as 1-2 doses of single agent ara-C or few doses of sorafenib are also allowed.
* Women of childbearing potential must practice contraception. Women considered not of childbearing potential include any of the following: no menses for at least 2 years or menses within 2 years but amenorrheic for at least 2 months and luteinizing hormone (LH) and follicular stimulating hormone (FSH) values within normal range (according to definition of postmenopausal for laboratory used) or bilateral oophorectomy or radiation castration and amenorrheic for at least 3 months. Females of childbearing potential should practice effective methods of contraception. Effective methods of contraception include barrier methods (e.g., condoms, diaphragm), spermicidal jelly or foam, oral, depo provera, or injectable contraceptives, intrauterine devices, tubal ligation, and abstinence. Male patients with female partners who are of childbearing potential should also practice contraception.
* Negative urine or serum pregnancy test.

Exclusion Criteria:

* Patients with known allergy or hypersensitivity to quizartinib, mannitol, AZA, cytarabine or any of their components.
* Serum potassium < 3.5 mEq/L despite supplementation, or > 5.5 mEq/L.
* Serum magnesium above or below the institutional normal limit despite adequate management.
* Serum calcium (corrected for albumin levels) above or below institutional normal limit despite adequate management.
* Patients with known significant impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of quizartinib.
* Patients with any other known disease concurrent severe and/or uncontrolled medical condition (e.g. uncontrolled diabetes, cardiovascular disease including congestive heart failure, myocardial infarction within 6 months and poorly controlled hypertension, chronic renal disease, or active uncontrolled infection) which could compromise participation in the study. Patients with current active malignancies or any remission for < 6 months, except patients with carcinoma in situ or with non-melanoma skin cancer who may have active disease or be in remission for less than 6 months.
* Patients with a known confirmed diagnosis of human immunodeficiency virus (HIV) infection or active viral hepatitis.
* Patients who have had any major surgical procedure within 14 days of day 1.
* Patients with known malignant disease of the central nervous system.
* Impaired cardiac function including any of the following: screening electrocardiography (ECG) with a corrected QT (QTc) > 450 msec. The QTc interval will be calculated by Fridericia's correction factor (QTcF) at screening and on day 5 prior to the first dose of AC220. The QTcF will be derived from the average QTcF in triplicate; if QTcF > 450 msec on day 5, AC220 will not be given; patients with congenital long QT syndrome; history or presence of sustained ventricular tachycardia requiring medical intervention; any history of clinically significant ventricular fibrillation or torsades de pointes; Known history of second or third degree heart block (may be eligible if the patient currently has a pacemaker); sustained heart rate of < 50/minute on pre-entry ECG; right bundle branch block + left anterior hemiblock (bifascicular block); patients with myocardial infarction or unstable angina within 6 months prior to starting study drug; congestive heart failure (CHF) New York (NY) Heart Association class III or IV. Atrial fibrillation documented within 2 weeks prior to first dose of study drug; patients who require treatment with concomitant drugs that prolong QT/QTc interval or strong CYP3A4 inhibitors or inducers with the exception of antibiotics, antifungals, and antivirals that are used as standard of care to prevent or treat infections and other such drugs that are considered absolutely essential for the care of the subject.
* Known family history of congenital long QT syndrome.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2013-11-12 (Actual); Primary Completion 2023-02-07 (Actual); Study Completion 2023-02-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yesid Alvarado, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Phase 1 Arm I (Quizartinib, Azacitidine) | Phase 1 Arm II (Quizartinib, Cytarabine) | Phase 2 Arm I (Quizartinib, Azacitidine) | Phase 2 Arm II (Quizartinib, Cytarabine)
Started | 5 | 1 | 35 | 32
Completed | 5 | 1 | 35 | 32
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase 1 Arm I (Quizartinib, Azacitidine) | Phase 1 Arm II (Quizartinib, Cytarabine) | Phase 2 Arm I (Quizartinib, Azacitidine) | Phase 2 Arm II (Quizartinib, Cytarabine) | Total
Number analyzed (Participants) | 5 | 1 | 35 | 32 | 73
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 1 | 14 | 7 | 25
  >=65 years | 2 | 0 | 21 | 25 | 48
Age, Continuous [Median (Full Range); unit: Years] | 47 [27 to 76] | 58 [58 to 58] | 68 [23 to 83] | 71 [55 to 84] | 69 [23 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 16 | 14 | 32
  Male | 3 | 1 | 19 | 18 | 41
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 4 | 1 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 3 | 2 | 5
  White | 3 | 1 | 26 | 29 | 59
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 2 | 0 | 3
Region of Enrollment [Number; unit: participants]
  United States | 5 | 1 | 35 | 32 | 73

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose of Quizartinib (Phase I)
Time Frame: At 28 days
Measure: Number; unit: Milligrams
Arm/Group | Phase 1 Arm I (Quizartinib, Azacitidine) | Phase 1 Arm II (Quizartinib, Cytarabine)
Number analyzed (Participants) | 5 | 1
Milligrams | 60 | 60

2. Primary Outcome: Participants With a Response
Description: (complete remission [CR]+complete response with incomplete bone marrow recovery [CRI]+partial remission [PR]+ hematologic improvement [HI]). Complete Rmission (CR) is bone marrow blasts of </= 5%, platelets >/= 100 and Absolute Neutrophil Count of >/= 1000. complete response with incomplete bone marrow recovery [CRI] is is bone marrow blasts of </= 5%, platelets >/= 100 or Absolute Neutrophil Count of >/= 1000. Hematologic improvement [HI]) is Bone Marrow Blasts </= 5%. Partial remission [PR] is bone marrow blasts of </= 5% with > 50% reduction, platelets >/= 100 and Absolute Neutrophil Count of >/= 1000.
Time Frame: At 56 days
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1 Arm I (Quizartinib, Azacitidine) | Phase 1 Arm II (Quizartinib, Cytarabine) | Phase 2 Arm I (Quizartinib, Azacitidine) | Phase 2 Arm II (Quizartinib, Cytarabine)
Number analyzed (Participants) | 5 | 1 | 35 | 32
Participants | 2 | 1 | 27 | 19

ADVERSE EVENTS:
Time Frame: Up to 9 years, 2 months
Arm/Group | Phase 1 Arm I (Quizartinib, Azacitidine) | Phase 1 Arm II (Quizartinib, Cytarabine) | Phase 2 Arm I (Quizartinib, Azacitidine) | Phase 2 Arm II (Quizartinib, Cytarabine)
All-Cause Mortality (participants affected / at risk) | 1/5 | 0/1 | 3/35 | 1/32
Serious Adverse Events (participants affected / at risk) | 1/5 | 0/1 | 14/35 | 21/32
Other Adverse Events (participants affected / at risk) | 5/5 | 1/1 | 32/35 | 32/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1 Arm I (Quizartinib, Azacitidine) (N=5) | Phase 1 Arm II (Quizartinib, Cytarabine) (N=1) | Phase 2 Arm I (Quizartinib, Azacitidine) (N=35) | Phase 2 Arm II (Quizartinib, Cytarabine) (N=32)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
Cardiac Arrest (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Death (General disorders) | 0 (0) | 0 (0) | 0 (0) | 5 (5)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Failure to Thrive (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Febrile Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 4 (4)
Fever (General disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Gastric Hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 2 (2) | 4 (5)
Colon Graft Versus Host Disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 0 (0) | 6 (6) | 3 (3)
Intracranial hemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Loss of peripheral Eye Sight (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 1 (1) | 0 (0) | 4 (6) | 9 (11)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (3)
Penumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash pustular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rectal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rectal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 1 (2)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Stroke (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thromboembolic event (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Transient ischemic attacks (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1 Arm I (Quizartinib, Azacitidine) (N=5) | Phase 1 Arm II (Quizartinib, Cytarabine) (N=1) | Phase 2 Arm I (Quizartinib, Azacitidine) (N=35) | Phase 2 Arm II (Quizartinib, Cytarabine) (N=32)
Black Hairy Tongue (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute Kidney Injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 5 (5)
Agitation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Alanine aminotransferase increased (Investigations) | 4 (4) | 1 (1) | 20 (20) | 11 (11)
Alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Allergic Rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1) | 4 (4)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 4 (4) | 6 (6)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 5 (7) | 7 (7)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Blood bilirubin increased (Investigations) | 4 (4) | 1 (1) | 20 (20) | 7 (7)
Bruising (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 3 (3)
Chest Pain (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Chills (General disorders) | 2 (2) | 0 (0) | 0 (0) | 4 (4)
Confusion (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 5 (5)
Conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 4 (4) | 5 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 4 (4) | 6 (6)
Creatinine decreased (Investigations) | 1 (2) | 0 (0) | 22 (23) | 5 (5)
Deconditioning (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Delirium (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 1 (1) | 6 (6) | 13 (13)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 3 (3) | 5 (5)
Dry eye (Eye disorders) | 3 (3) | 0 (0) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 6 (6)
Edema (General disorders) | 3 (3) | 0 (0) | 2 (2) | 6 (8)
Electrocardiogram QT corrected interval prolonged (Investigations) | 1 (1) | 0 (0) | 4 (4) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 4 (4)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 6 (6)
Fatigue (General disorders) | 1 (1) | 1 (1) | 8 (8) | 8 (8)
Febrile neutropenia (Blood and lymphatic system disorders) | 3 (3) | 1 (2) | 14 (18) | 8 (9)
Fever (General disorders) | 1 (1) | 0 (0) | 2 (3) | 5 (5)
Flu like symptoms (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
fluid overload (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 2 (2) | 0 (0) | 2 (2) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 4 (4) | 4 (4)
Gum bleeding (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hallucinations (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Headache (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 4 (5)
Hematoma (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hemorrhage (General disorders) | 0 (0) | 0 (0) | 3 (3) | 5 (5)
Hemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 7 (9) | 6 (6)
Hypermagnesemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 3 (3) | 2 (2)
Hypernatremia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 4 (4) | 2 (2)
Hyperphosphatemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 7 (7) | 5 (5)
Hyperuricemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 6 (6) | 7 (7)
Hypocalcemia (Metabolism and nutrition disorders) | 4 (5) | 1 (1) | 20 (20) | 9 (9)
Hypokalemia (Metabolism and nutrition disorders) | 4 (4) | 1 (1) | 22 (22) | 9 (9)
Hypomagnesemia (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (1) | 23 (23) | 9 (9)
Hyponatremia (Metabolism and nutrition disorders) | 3 (3) | 1 (1) | 15 (15) | 8 (8)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 11 (11) | 2 (2)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 3 (3) | 9 (9)
Infection (Infections and infestations) | 2 (3) | 0 (0) | 11 (13) | 8 (9)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Lung infection (Infections and infestations) | 2 (2) | 1 (1) | 6 (6) | 12 (15)
Malaise (General disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
mouth sores (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 5 (5)
Mucositis oral (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2) | 4 (4)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Nausea (Gastrointestinal disorders) | 3 (3) | 0 (0) | 8 (9) | 14 (14)
Neutrophil count decreased (Investigations) | 2 (2) | 0 (0) | 1 (1) | 9 (9)
Pain (General disorders) | 3 (7) | 0 (0) | 7 (12) | 16 (35)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Phosphorus increased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Platelet count decreased (Investigations) | 2 (2) | 1 (1) | 3 (3) | 8 (8)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (2) | 3 (3)
Pneumonitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 9 (9)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 3 (3) | 2 (2)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 5 (5)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Ulcer (General disorders) | 1 (2) | 0 (0) | 0 (0) | 2 (4)
Hyperuricemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 5 (5) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 5 (5)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0) | 5 (5) | 9 (9)
White blood cell decreased (Investigations) | 1 (1) | 1 (1) | 2 (2) | 13 (13)
wound (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-02-25): https://cdn.clinicaltrials.gov/large-docs/71/NCT01892371/Prot_SAP_000.pdf